CLINICAL TRIAL: NCT00896493
Title: A Phase II Study of Non-myeloablative Allogeneic Transplantation Using Total Lymphoid Irradiation (TLI) and Antithymocyte Globulin (ATG) In Patients With Cutaneous T Cell Lymphoma
Brief Title: Ph II of Non-myeloablative Allogeneic Transplantation Using TLI & ATG In Patients w/ Cutaneous T Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Wen-Kai Weng, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-16213; SU-04062009-2138 (Other: Stanford University); 16213 (Other: Stanford IRB); BMT206 (Other: OnCore)
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Results first posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Mycoses; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous; Bone Marrow Transplant Failure; Lymphoma, Non-Hodgkin; Cutaneous T-cell Lymphoma
MeSH Terms: conditions — Mycoses; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous; Lymphoma, Non-Hodgkin | interventions — Antilymphocyte Serum; Cyclosporine; Lymphatic Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Total lymphoid irradiation & anti-thymocyte immunoglobulin (Experimental): TLI is administered from a 6 MeV linear accelerator in 80c- 120c Gy fractions. Anti-thymocyte-Globulin (ATG) is administered intravenously for a total dose of 7.5 mg/kg.
  Interventions: Drug: anti-thymocyte globulin; Drug: cyclosporine; Radiation: Lymphoid radiation

INTERVENTIONS:
Drug: anti-thymocyte globulin — ATG will be administered five times intravenously at 1.5 mg/kg/day from day -11 through day -7 for a total dose of 7.5 mg/kg
  Other Names: ATG
Drug: cyclosporine — 5 mg/kg PO or IV
  Other Names: cyclosporin; cyclosporin A
Radiation: Lymphoid radiation — TLI is administered ten times in 80c- 120c Gy fractions on day -11 through day -7 and day -4 through day -1
  Other Names: Total lymphoid irradiation (TLI)

SUMMARY:
Non-myeloablative approach for allogeneic transplant is a reasonable option, especially given that the median age at diagnosis is 55-60 years and frequently present compromised skin in these patients, which increases the risk of infection. Therefore, we propose a clinical study with allogeneic hematopoietic stem cell transplantation (HSCT) using a unique non-myeloablative preparative regimen, TLI/ATG, to treat advanced mycosis fungoides/Sezary syndrome (MF/SS).

DETAILED DESCRIPTION:
Primary Objectives

-To evaluate the graft versus lymphoma effect by monitoring rate of clinical response, event-free and overall survival.

Secondary Objectives

-To evaluate the incidence and extent of acute and chronic graft-versus-host disease (GVHD) and time to engraftment.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IIB-IV mycosis fungoides or Sezary syndrome, who have failed at least 1 standard systemic therapy or are not candidates for standard therapy.
2. Pathology reviewed and the diagnosis confirmed at Stanford University Medical Center.
3. Age > 18 years and <= 75 years.
4. Karnofsky Performance Status >= 70%.
5. Corrected DLCO >= 40%
6. Left ventricle ejection fraction (LVEF) > 30%.
7. ALT and AST must be <= 3X normal. Total bilirubin <= 3 mg/dL unless hemolysis or Gilbert's disease.
8. Estimated creatinine clearance >= 50 ml/min.
9. Have a related or unrelated HLA-identical donor or one antigen/allele mismatched in HLA-A, B, C or DRB1.
10. Signed informed consent.
11. Patients with prior malignancies diagnosed > 5 years ago without evidence of disease are eligible.
12. Patients with a prior malignancy treated < 5 years ago but have a life expectancy of > 5 years for that malignancy are eligible.

Donor Inclusion Criteria

1. Age >=17.
2. HIV seronegative.
3. No contraindication to the administration of G-CSF.
4. Willing to have a central venous catheter placed for apheresis if peripheral veins are inadequate

Exclusion Criteria:

1. Uncontrolled active infection.
2. Uncontrolled congestive heart failure or angina.
3. Pregnancy or nursing patients will be excluded from the study.
4. Those who are HIV-positive will be excluded from the study due to high risk of lethal infection after hematopoietic cell transplantation.

Donor Exclusion Criteria

1. Serious medical or psychological illness.
2. Pregnant or lactating women are not eligible
3. Prior malignancies within the last 5 years except for non-melanoma skin cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-05; Primary Completion 2021-11-06 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Kai Weng, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jagasia MH, Greinix HT, Arora M, Williams KM, Wolff D, Cowen EW, Palmer J, Weisdorf D, Treister NS, Cheng GS, Kerr H, Stratton P, Duarte RF, McDonald GB, Inamoto Y, Vigorito A, Arai S, Datiles MB, Jacobsohn D, Heller T, Kitko CL, Mitchell SA, Martin PJ, Shulman H, Wu RS, Cutler CS, Vogelsang GB, Lee SJ, Pavletic SZ, Flowers ME. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant. 2015 Mar;21(3):389-401.e1. doi: 10.1016/j.bbmt.2014.12.001. Epub 2014 Dec 18. PMID 25529383
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Result] Weng WK, Arai S, Rezvani A, Johnston L, Lowsky R, Miklos D, Shizuru J, Muffly L, Meyer E, Negrin RS, Wang E, Almazan T, Million L, Khodadoust M, Li S, Hoppe RT, Kim YH. Nonmyeloablative allogeneic transplantation achieves clinical and molecular remission in cutaneous T-cell lymphoma. Blood Adv. 2020 Sep 22;4(18):4474-4482. doi: 10.1182/bloodadvances.2020001627. PMID 32941647
- [Derived] Weng WK, Armstrong R, Arai S, Desmarais C, Hoppe R, Kim YH. Minimal residual disease monitoring with high-throughput sequencing of T cell receptors in cutaneous T cell lymphoma. Sci Transl Med. 2013 Dec 4;5(214):214ra171. doi: 10.1126/scitranslmed.3007420. PMID 24307695

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin: Total lymphoid irradiation (TLI) is administered from a 6 MeV linear accelerator in 80c- 120c Gy fractions. Anti-thymocyte-Globulin (ATG) is administered intravenously for a total dose of 7.5 mg/kg.
Period: Overall Study
Arm/Group | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin
Started | 38
Completed Assigned Treatment | 35
Completed | 35
Not Completed | 3
Not completed — Early disease relapse | 3

BASELINE CHARACTERISTICS:
Arm/Group | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 62 [20 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 31
  Black | 4
  Asian | 2
  Unknown/not reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38
Diagnosis [Count of Participants; unit: Participants]
  Mycosis fungoides | 20
  Sezary Syndrome | 18
Retro-CLIPI [Count of Participants; unit: Participants] — Risk stratification using the Retrospective Cutaneous Lymphoma International Prognostic Index (Retro-CLIPI). Population: Participants who completed assigned treatment
  Participants
    High risk: number analyzed (Participants) | 35
    High risk | 18
    Intermediate risk: number analyzed (Participants) | 35
    Intermediate risk | 13
    Low risk: number analyzed (Participants) | 35
    Low risk | 4
Time from diagnosis to allogeneic HCT [Median (Full Range); unit: months] — HCT: hematopoietic cell transplantation Population: Participants who completed assigned treatment
  months
    number analyzed (Participants) | 35
    (all) | 40 [9 to 152]
Active disease at the time of conditioning [Count of Participants; unit: Participants] — Participants may have had more than one active disease Population: Participants who completed assigned treatment
  Participants
    Skin: number analyzed (Participants) | 35
    Skin | 35
    Blood: number analyzed (Participants) | 35
    Blood | 12
    Lymph node: number analyzed (Participants) | 35
    Lymph node | 22
    Visceral (site: bone marrow): number analyzed (Participants) | 35
    Visceral (site: bone marrow) | 4
    Visceral (site: tonsil): number analyzed (Participants) | 35
    Visceral (site: tonsil) | 1
Donor [Count of Participants; unit: Participants] — Population: Participants who completed assigned treatment
  Participants
    Sibling: number analyzed (Participants) | 35
    Sibling | 13
    Unrelated - matched: number analyzed (Participants) | 35
    Unrelated - matched | 15
    Unrelated - unmatched: number analyzed (Participants) | 35
    Unrelated - unmatched | 7
Donor-recipient cytomegalovirus (CMV) status [Count of Participants; unit: Participants] — Population: Participants who completed assigned treatment
  Participants
    Donor and/or recipient seropositive: number analyzed (Participants) | 35
    Donor and/or recipient seropositive | 27
    Donor and recipient seronegative: number analyzed (Participants) | 35
    Donor and recipient seronegative | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) at 180 Days
Description: Progression-Free Survival (PFS; time to disease progression or death from any cause) assessed at 180 days (Kaplan-Meier estimate). Disease progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 180 days
Population: Participants who completed assigned treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin
Number analyzed (Participants) | 35
percentage of participants | 73 [55 to 85]

2. Secondary Outcome: Number of Participants With Acute Graft-versus-host Disease (GVHD)
Description: Cumulative incidence at 6 months. GvHD was assessed using the 2015 NIH consensus criteria.
Time Frame: 6 months
Population: Participants who completed assigned treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin
Number analyzed (Participants) | 35
Participants
  Any Grade | 9
  Grade II-IV | 5

3. Secondary Outcome: Number of Participants With Chronic Graft-versus-host Disease (GVHD)
Description: Cumulative incidence at 6 months (any grade). GvHD was assessed using the 2015 NIH consensus criteria.
Time Frame: 2 years
Population: Participants who completed assigned treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin
Number analyzed (Participants) | 35
Participants | 9

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is the time measurement between the day of allogeneic transplant and death from any cause (Kaplan-Meier estimate).
Time Frame: 2 years
Population: Participants who completed assigned treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin
Number analyzed (Participants) | 35
percentage of participants | 68 [50 to 81]

5. Secondary Outcome: Overall Survival (OS)
Description: as for outcome 4
Time Frame: 5 years
Population: Participants who completed assigned treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin
Number analyzed (Participants) | 35
percentage of participants | 56 [38 to 71]

6. Secondary Outcome: Mortality
Description: Total count of non-relapsed mortality and mortality from relapsed disease.
Time Frame: Up to 5 years
Population: Participants who completed assigned treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin
Number analyzed (Participants) | 35
Participants
  Non-relaped, treatment related | 5
  Non-relaped, not treatment related | 1
  Disease relapse | 15

7. Secondary Outcome: Treatment Related Mortality
Time Frame: Up to 5 years
Population: Participants who completed assigned treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin
Number analyzed (Participants) | 35
Participants
  Acute GVHD | 1
  Chronic GVHD | 1
  Secondary malignancy | 1
  Hepatitis B | 1
  Hemorrhage secondary to anticoagulation | 1

8. Secondary Outcome: Event Free Survival (EFS)
Description: Event-free survival (EFS) is the time measurement between the day of allogeneic transplant and the first documented recurrence or death from any cause (Kaplan-Meier estimate).
Time Frame: 2 years
Population: Participants who completed assigned treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin
Number analyzed (Participants) | 35
percentage of participants | 40 [24 to 56]

9. Secondary Outcome: Event Free Survival (EFS)
Description: as for outcome 8
Time Frame: 5 years
Population: Participants who completed assigned treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin
Number analyzed (Participants) | 35
percentage of participants | 26 [13 to 41]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin
All-Cause Mortality (participants affected / at risk) | 21/38
Serious Adverse Events (participants affected / at risk) | 7/38
Other Adverse Events (participants affected / at risk) | 20/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin (N=38)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Acute lymphoblastic leukemia
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Metastatic cutaneous squamous cell carcinoma
Acute Viral Hepatitis (Hepatobiliary disorders) | 1 — Hepatitis B infection
Liver Failure (Hepatobiliary disorders) | 1 — Liver failure due to disease progression
Sepsis (Infections and infestations) | 1
GI Bleeding (Gastrointestinal disorders) | 1 — Acute GI GVHD
Hyperbilirubinemia (Hepatobiliary disorders) | 1 — Acute Liver GVHD
Multi-organ failure (General disorders) | 1 — Secondary to acute GVHD
Acute appendicitis (Gastrointestinal disorders) | 1
Hemorrhage (General disorders) | 1 — Internal bleeding from anti-coagulation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Lymphoid Irradiation & Anti-thymocyte Immunoglobulin (N=38)
Serum sickness (Injury, poisoning and procedural complications) | 3 — Serum sickness from ATG infusion
Disease Relapse (General disorders) | 20 — Relapse of lymphoma
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 — Localized cutaneous squamous cell carcinoma
Anemia (Blood and lymphatic system disorders) | 16 — Anemia needing transfusion
Neutropenia (Blood and lymphatic system disorders) | 6 — Neutrophil <0.5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 — Platelet count <10,000
Neutropenic fever (Infections and infestations) | 3
Infection, non-specified (Infections and infestations) | 4 — Central-line related infection
Vaginal bleeding (Reproductive system and breast disorders) | 1
Post transplant lymphoproliferative disorder (PTLD) (Infections and infestations) | 2 — Post-transplant lymphoproliferative disorder (PTLD) secondary to Epstein Barr virus (EBV) reactivation
CMV viremia (Infections and infestations) | 17
EBV viremia (Infections and infestations) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT00896493/Prot_SAP_001.pdf
  • Informed Consent Form (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT00896493/ICF_000.pdf